CLINICAL TRIAL: NCT00059371
Title: Trial of Male Circumcision to Reduce HIV Incidence
Brief Title: Male Circumcision and HIV Rates in Kenya
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Carolyn Williams, Chief Epidemiology, NIAID
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 5U01AI050440-02 (NIH)
Record Dates: First submitted 2003-04-23; First posted 2003-04-24 (Estimated); Last update posted 2008-05-30 (Estimated); Status verified 2007-09

CONDITIONS: HIV Infections
Keywords: Male circumcision; HIV acquisition; Sexually transmitted infection; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases | interventions — Circumcision, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Circumcised immediately (Active Comparator)
  Interventions: Procedure: male circumcision
- Delayed Circumcision (Placebo Comparator): Men who were randomized to delayed circumcision were scheduled to be offered male circumcision 2 years after their randomization.
  Interventions: Procedure: male circumcision

INTERVENTIONS:
Procedure: male circumcision

SUMMARY:
The Luo tribe of Kisumu, Kenya, does not traditionally practice male circumcision (MC). This study will work with the Luo tribe to test the effectiveness of MC on reducing the risk of HIV infections in young men.

DETAILED DESCRIPTION:
Since 1989, numerous epidemiological studies have reported a significant association between lack of male circumcision (MC) and risk for HIV infection through heterosexual intercourse. These results have led to calls for male circumcision to be considered as an additional HIV prevention strategy. However, there is a consensus among the international health community that a randomized controlled trial of MC is needed to control for possible confounding factors. Additionally, known risks associated with MC need further investigation. This study will assess the effectiveness of male circumcision in reducing HIV incidence and will evaluate complications of the MC procedure, changes in sexual behavior following circumcision, and the biological mechanisms by which the foreskin may increase HIV susceptibility. The study will be conducted in Kisumu, Kenya, where the Luo tribe is the main ethnic group and less than 10% of adult men are circumcised.

Uncircumcised men aged 18 to 24 years old will be offered voluntary HIV counseling and testing. HIV negative men will be asked to enroll in the study. All study participants will be interviewed to obtain socio-demographic information and assess behavioral risk factors. Participants will be examined for significant medical conditions. All men will be counseled in strategies to reduce their risk for HIV infection. Consenting men will be randomly assigned to either the treatment (circumcised) arm or the control (uncircumcised) arm of the study. After circumcision, men will be monitored for complications. They will be counseled to abstain from sex until healing is complete. Follow-up visits will occur every 6 months for 2 years. Uncircumcised men will be offered circumcision at the end of follow-up.

The primary study endpoints will be HIV incidence and surgical complications. Additional outcomes will be the incidence of other sexually transmitted diseases and behavioral risks. Additional laboratory studies of foreskin tissue will evaluate the number and density of specialized cells rich in HIV receptors in order to illuminate the biological mechanisms by which presence of foreskin may increase HIV susceptibility.

ELIGIBILITY:
Inclusion Criteria

* HIV uninfected and willing to be tested
* Live in Kisumu District, Kenya
* Uncircumcised but willing to be circumcised
* At least one sexual partner in the 12 months prior to study entry

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2887 (Actual)
Dates: Start 2002-02; Primary Completion 2006-10 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
HIV incidence | 2 years
surgical complications | 2 years

SECONDARY OUTCOMES:
incidence of other sexually transmitted diseases | 2 years
behavioral risks | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Bailey, PhD, MPH, Principal Investigator — University of Illinois at Chicago
Locations (1):
- UNIM Clinic, Kisumu, Kisumu County, Kenya

REFERENCES:
- [Derived] Davis SM, Pals S, Yang C, Odoyo-June E, Chang J, Walters MS, Jaoko W, Bock N, Westerman L, Toledo C, Bailey RC. Circumcision status at HIV infection is not associated with plasma viral load in men: analysis of specimens from a randomized controlled trial. BMC Infect Dis. 2018 Jul 28;18(1):350. doi: 10.1186/s12879-018-3257-8. PMID 30055581
- [Derived] Mehta SD, Gaydos C, Maclean I, Odoyo-June E, Moses S, Agunda L, Quinn N, Bailey RC. The effect of medical male circumcision on urogenital Mycoplasma genitalium among men in Kisumu, Kenya. Sex Transm Dis. 2012 Apr;39(4):276-80. doi: 10.1097/OLQ.0b013e318240189c. PMID 22421693
- [Derived] Mehta SD, Maclean I, Ndinya-Achola JO, Moses S, Martin I, Ronald A, Agunda L, Murugu R, Bailey RC, Melendez J, Zenilman JM. Emergence of quinolone resistance and cephalosporin MIC creep in Neisseria gonorrhoeae isolates from a cohort of young men in Kisumu, Kenya, 2002 to 2009. Antimicrob Agents Chemother. 2011 Aug;55(8):3882-8. doi: 10.1128/AAC.00155-11. Epub 2011 May 23. PMID 21606224
- [Derived] Mehta SD, Gray RH, Auvert B, Moses S, Kigozi G, Taljaard D, Puren A, Agot K, Serwadda D, Parker CB, Wawer MJ, Bailey RC. Does sex in the early period after circumcision increase HIV-seroconversion risk? Pooled analysis of adult male circumcision clinical trials. AIDS. 2009 Jul 31;23(12):1557-64. doi: 10.1097/QAD.0b013e32832afe95. PMID 19571722
- [Derived] Bailey RC, Moses S, Parker CB, Agot K, Maclean I, Krieger JN, Williams CF, Campbell RT, Ndinya-Achola JO. Male circumcision for HIV prevention in young men in Kisumu, Kenya: a randomised controlled trial. Lancet. 2007 Feb 24;369(9562):643-56. doi: 10.1016/S0140-6736(07)60312-2. PMID 17321310